CLINICAL TRIAL: NCT05252520
Title: A Phase 1 Open-label Single Ascending Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of JNJ-77474462 (Bermekimab) in Healthy Chinese Participants Following Subcutaneous Administration
Brief Title: A Study of JNJ-77474462 (Bermekimab) in Healthy Chinese Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The development of bermekimab in Immunology is stopped
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR109109; 77474462HDS1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-02-16; First posted 2022-02-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — bermekimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-77474462 (Experimental): Participants will receive a single subcutaneous (SC) Dose 1 of JNJ-77474462 on Day 1 in Cohort 1, a single SC Dose 2 of JNJ-77474462 on Day 1 in Cohort 2 and a single SC Dose 3 of JNJ-77474462 on Day 1 in Cohort 3.
  Interventions: Drug: JNJ-77474462

INTERVENTIONS:
Drug: JNJ-77474462 — JNJ-77474462 will be administered subcutaneously.
  Other Names: Bermekimab

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of JNJ-77474462 following single ascending dose subcutaneous (SC) administration to healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 27.9 kilograms per meter square (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of between 50 to 90 kg, inclusive
* Otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and Day -2 to -1. Any abnormalities must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* A female of childbearing potential must have a negative pregnancy test at screening and on Day -2 to -1
* Must have 3 quadrants on the abdomen where the skin is not tender, bruised, red, scaly, hardened, or tattooed for subcutaneous (SC) administration
* Must be a nonsmoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, endocrine, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 12 months before Screening or positive test result(s) for alcohol or drugs of abuse (including morphine, ketamine, tetrahydrocannabinolic acid, methamphetamine, dimethylene dioxoamphetamine, cocaine) at Screening and Day -2 to -1
* Have a history of active granulomatous infection (including histoplasmosis or coccidioidomycosis), nontuberculous mycobacterial infection or opportunistic infection (including pneumocystosis, aspergillosis, and disseminated herpes zoster defined as zoster with central nervous system involvement or zoster spreading to more than 2 adjacent dermatomes)
* Has a chest radiograph within 3 months before the first administration of study intervention that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis (TB). A chest computerized tomography (CT) scan is also acceptable if already available or obtained outside of the study protocol
* Has tested positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and treponema pallidum-specific antibody

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of JNJ-77474462 | Up to Day 85
  Cmax is defined as the maximum observed serum concentration of JNJ-77474462.
Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-77474462 | Up to Day 85
  Tmax is defined as the time to reach maximum observed serum concentration of JNJ-77474462.
Area Under the Serum Concentration Versus Time Curve from Time Zero to Infinity (AUC [0-Infinity]) of JNJ-77474462 | Up to Day 85
  AUC (0-infinity) is defined as the area under the serum concentration of JNJ-77474462 versus time curve from time zero to infinity with extrapolation of the terminal phase.
Area Under the Serum Concentration Versus Time Curve from Time Zero to the Time Corresponding to the Last Quantifiable Concentration (AUC [0-Last]) of JNJ-77474462 | Up to Day 85
  AUC (0-Last) is defined as the area under the serum concentration of JNJ-77474462 versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Terminal Half-life (T1/2) of JNJ-77474462 | Up to Day 85
  T1/2 will be reported. T1/2 is defined as the terminal half-life of JNJ-77474462.
Apparent Total Systemic Clearance after Extravascular Administration (CL/F) of JNJ-77474462 | Up to Day 85
  CL/F is defined as the apparent total systemic clearance after extravascular administration of JNJ-77474462.
Apparent Volume of Distribution Based on Terminal Phase After Extravascular Administration (Vz/F) of JNJ-77474462 | Up to Day 85
  Vz/F is defined as the apparent volume of distribution based on terminal phase after extravascular administration of JNJ-77474462.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) by Severity | Up to Day 85
  Percentage of participants with TEAEs by severity will be reported. An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study intervention through Day 85 is considered to be treatment-emergent. Severity will be assessed based on the following categories: a) Mild: Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities, b) Moderate: Sufficient discomfort is present to cause interference with normal activity and c) Severe: Extreme distress, causing significant impairment of functioning or incapacitation. Prevents normal everyday activities.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Day 85
  Percentage of participants with SAEs will be reported. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important to prevent one of the outcomes listed above.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 85
  Number of participants with clinically significant changes in vital signs (temperature, pulse/heart rate, respiratory rate and blood pressure) will be reported.
Number of Participants with Clinically Significant Changes in Electrocardiograms (ECGs) | Up to Day 85
  Number of participants with clinically significant changes in ECGs will be reported.
Number of Participants with Clinically Significant Changes in Hematology Parameters | Up to Day 85
  Number of participants with clinically significant changes in hematology parameters will be reported.
Number of Participants with Clinically Significant Changes in Chemistry Parameters | Up to Day 85
  Number of participants with clinically significant changes in chemistry parameters will be reported.
Number of Participants with Clinically Significant Changes in Urinalysis | Up to Day 85
  Number of participants with clinically significant changes in urinalysis will be reported.
Number of Participants with Presence of Antibodies to JNJ-77474462 | Up to Day 85
  Number of participants with presence of antibodies to JNJ-77474462 will be reported. The detection and characterization of antibodies to JNJ-77474462 will be performed using a validated drug-tolerant method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://www.janssen.com/clinical-trials/transparency